CLINICAL TRIAL: NCT04445428
Title: Oral Polio Vaccine as Potential Protection Against COVID-19: A Cluster-randomised Trial in Guinea-Bissau
Brief Title: OPV as Potential Protection Against COVID-19
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bandim Health Project (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 77/CNES/INASA/2020
Record Dates: First submitted 2020-06-22; First posted 2020-06-24 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Poliovirus Vaccine, Oral; COVID; Mortality; Morbidity; Non-Specific Effects of Vaccines
MeSH Terms: interventions — Poliovirus Vaccine, Oral

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Participants are cluster randomised to OPV or no vaccine. Information on group assignment is not available to health center staff and staff at the health and demographic surveillance system
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Standard dose bivalent oral polio vaccine, 0.1ml, and information regarding prevention of COVID-19
  Interventions: Biological: oral polio vaccine + information; Behavioral: Information
- Control (Other): Information regarding prevention of COVID-19
  Interventions: Behavioral: Information

INTERVENTIONS:
Biological: oral polio vaccine + information — Bivalent OPV (GSK), 0.1 ml administered orally on a sugar lump
  Arms: Intervention
Behavioral: Information — Advice regarding how to protect oneself from COVID-19

SUMMARY:
Since the 1960s, studies have shown that oral polio vaccine (OPV) may have beneficial non-specific effects, reducing morbidity and mortality from other infections than polio. Such beneficial non-specific effect have been observed for other live vaccines, including measles, smallpox and BCG vaccine. For BCG, the vaccine for which the mechanism has been studied the most, the effects appear to be mediated through the innate immune system. The COVID-19 pandemic caused by the novel coronavirus SARS-CoV-2 has now caused over 7.1 million cases and >400,000 deaths worldwide. As everywhere else, it is anticipated that in Africa the older part of the population will be at risk of severe COVID-19. OPV is widely used in Africa, but for children. Both polio and coronavirus are positive-strand RNA viruses, therefore it is likely that they may induce and be affected by common innate immune mechanisms.

In a randomised trial at the Bandim Health Project in Guinea-Bissau, the investigators will assess the effect of providing OPV vs no vaccine to 3400 persons above 50 years of age. The trial will have the power to test the hypothesis that OPV reduces the combined risk of morbidity admission or death (composite outcome) by at least 28% over the subsequent 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Living in a household which has had a census visit conducted after 1 January in 2017. Age above 50.

Exclusion Criteria:

* Previous adverse events to OPV; Previous documented COVID-19; Acute severe infection.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3400 (Estimated)
Dates: Start 2020-07-15 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Mortality or infectious disease causing consultation or admission (Composite outcome) | 6 months
  Composite outcome of the first of death, hospitalisation for infection and/or consultation for infection at the health centre

SECONDARY OUTCOMES:
Self-reported morbidity | 6 months
  Episodes with self-reported infectious disease morbidity.
Suspected COVID-19 infection | 6 months
  Episodes with self-reported infectious disease morbidity suspected to be caused by COVID (three or more of the following: fever, cough, sore thought, extreme fatigue, loss of smell/taste).
Mortality | 6 months
  Either of the components of the composite outcome.
Hospital admission for infectious disease | 6 months
  Either of the components of the composite outcome included repeated events.
Consultations for infectious disease | 6 months
  Either of the components of the composite outcome included repeated events.

CONTACTS AND LOCATIONS:
Overall Officials: Ane Fisker, MD, PhD, Principal Investigator — Bandim Health Project
Locations (1):
- Bandim Health Project, Bissau, Guinea-Bissau

IPD SHARING:
Plan to Share IPD: No
Provided request, data can be made available

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-11-16): https://cdn.clinicaltrials.gov/large-docs/28/NCT04445428/SAP_000.pdf